CLINICAL TRIAL: NCT04059068
Title: Understanding the Role of Macrophage-mediated Inflammation in White Adipose Tissue and Liver Fibrosis
Brief Title: Macrophage-mediated Inflammation in White Adipose Tissue and Non-alcoholic Fatty Liver Disease.
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 19HH5303
Record Dates: First submitted 2019-08-15; First posted 2019-08-16 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: macrophage; adipose tissue; fibroblast; liver disease; RNA sequencing
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Adipose tissue (6-8g) Liver tissue (1g) Blood (10ml) The samples will be used for analysis specifically for RNA, protein or imaging. They will either be cryo-preserved or snap frozen to prevent them from perishing. They can be stored in liquid nitrogen or -80 deg Celcius freezer for up to 10 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- NASH (non-alcoholic steatohepatitis): Patients diagnosed with non-alcoholic steatohepatitis.
- NAFLD (non-alcoholic fatty liver disease): Patients diagnosed with non-alcoholic fatty liver disease.
- Control: Patients with normal liver tissue.
- obese / high WAT inflammation and fibrosis: Patients who are obese with inflammed white adipose tissue and evidence of fibrosis.
- obese / low WAT inflammation and fibrosis: Patients who are obese with no evidence of inflammed white adipose tissue and no evidence of fibrosis.
- non- obese controls: Patients who are not obese.

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is present in one third of the population and due to its potential to cause irreversible liver damage and liver cancer, it is a significant health burden. There is a strong link between obesity and NALFD. As fat accumulates, the body is unable to process it, leading to unhealthy fat metabolism. Currently, other than lifestyle measures and better control of Type 2 Diabetes Mellitus (T2DM) with medication, there is no drug that can prevent or reverse the liver damage. Furthermore, there is no easy way to identify which person will go on to develop the liver damage.

Mounting evidence suggests that inflammation in the fat has a key role in driving liver damage, particularly by the immune cell called the macrophage. However, detailed mechanisms are lacking. Therefore, the aim of this proposal is to study obese patients with NAFLD to better understand the link between unhealthy fat metabolism and liver damage, focusing on identifying macrophage-derived drug targets which can potentially reverse the liver disease. Samples of fat and liver from patients who are having bariatric surgery at Imperial College Healthcare NHS Trust will be analysed to identify and target the inflammatory markers of unhealthy fat and NAFLD using genetic profiling techniques.

DETAILED DESCRIPTION:
NAFLD is a huge health burden and can lead to liver damage,scarring and cancer, therefore gaining a further understanding of the mechanisms involved in causing liver damage is particularly important to identify drug targets that could reverse this process.

White adipose tissue (WAT) or fat fails to respond normally in obesity which leads to fat deposition in other organs, particularly the liver, and the fat tissue becomes inflamed. The inflammation in the fat is lead by specific immune cells called macrophages. This inflammatory state in the fat tissue is thought to be a precursor to liver inflammation and liver damage. This has been demonstrated in mouse models where the fat inflammatory cells contributed to liver inflammation and worsened liver damage, emphasising the importance of the relationship between fat tissue and the liver in NAFLD.

Liver damage or liver fibrosis is also the result of activation of these inflammatory cells, the macrophages, in the liver which drive scarring through cells called fibroblasts that lay down collagen. Therefore, understanding the interaction between the cells involved in inflammation (macrophages) and scarring (fibroblasts) in both the fat and the liver is key to identifying potential drug targets for reversal of this process.

|the investigators demonstrated, using an obese animal model, that the release of pro-fibrotic compounds called prostagladins from the fat macrophages is linked to NAFLD and liver inflammation. Based on these results the investigators aim to deepen the understanding of the link between fat and liver inflammation and damage specifically looking at cell interactions (the macrophage and fibroblast) by using genetic tests on liver and fat samples in obese participants.

ELIGIBILITY:
Inclusion Criteria:

* Bariatric and Upper Gastrointestinal (UGI) surgery patients classified as obese or morbidly obese (BMI >30)
* Patients who attend UGI cancer services with a BMI <25

Exclusion Criteria:

Participants with:

* alcohol consumption more than 10g of ethanol per day
* viral Hepatitis infection
* HIV
* Autoimmune condition
* genetic liver disease
* other metabolic causes of liver disease
* abnormal clotting
* immunosuppressive medication
* drugs that are known to precipitate hepatic steatosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are attending the bariatric services at St Mary hospital and UGI services at Hammersmith Hospital, Imperial College Healthcare NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Macrophage ligand-fibroblast receptor | 3 years
  Macrophage ligand-fibroblast receptors that are assessed by single cell-RNA-sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Behmoaras, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No